CLINICAL TRIAL: NCT07283302
Title: Pre-operative Rehabilitation Protocol for a Pediatric Patient With Humeral Head and Shaft Deformity: A Case Report
Brief Title: Pre-Surgery Rehab for a Child With Humeral Head and Shaft Deformity: A Case Report
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sameh Eldaly, Researcher, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/006101
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Osteomyelitis Chronic; Bone Defects
Keywords: Pre-operative rehabilitation; Humeral head deformity; Upper limb deformity; Pre-operative rehabilitation (prehabilitation)
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation; Low-Level Light Therapy; Musculoskeletal Manipulations; Phonophoresis; High-Energy Shock Waves; Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interventional (Experimental): This single-arm case report includes a structured pre-operative physical therapy rehabilitation program for a pediatric patient with humeral head and shaft deformity. The intervention consists of supervised sessions incorporating pain-modulation modalities (as clinically indicated), manual therapy to improve shoulder mobility, therapeutic exercises for flexibility, strengthening, and neuromuscular control, and scapular stabilization/positioning strategies (including taping as needed). Treatment is progressed based on tolerance and clinical response, with the goal of improving pre-operative shoulder pain, range of motion, strength, posture, and functional use of the upper limb.
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation; Device: Low-Level Laser Therapy; Other: Manual Therapy; Other: Phonophoresis; Other: PNF stretching; Other: kinesio taping

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation — a method of pain relief that uses a device to send low-voltage electrical impulses through electrodes placed on the skin
Device: Low-Level Laser Therapy — a non-invasive medical treatment that uses low-level lasers or light-emitting diodes (LEDs) to stimulate cell function and accelerate the body's natural healing process
Other: Manual Therapy — a hands-on treatment approach
Other: Phonophoresis — a medical procedure that uses therapeutic ultrasound to deliver topical medications through the skin and into deeper tissues
  Other Names: Ultrasound
Other: PNF stretching — is an advanced technique that combines muscle contraction and relaxation to increase flexibility and range of motion
Other: kinesio taping — Kinesio tape will be applied to the shoulder and scapular region to support improved alignment and scapular control during movement.

SUMMARY:
The goal of this observational study (single-patient case report) is to learn whether a structured pre-operative physical therapy rehabilitation program can improve shoulder function, reduce pain, and improve quality of life in an 11-year-old girl with humeral head and shaft deformity (post-inflammatory changes).

The main questions it aims to answer are:

Does shoulder range of motion and muscle strength improve after the program? Does pain and functional ability (including posture) improve after the program?

Participants will:

Attend 12 sessions over October-November 2025 (2 sessions/week) at the Faculty of Physical Therapy, Cairo University

Receive a standardized session program that may include:

TENS, low-level laser therapy, manual therapy (Spencer technique), phonophoresis PNF stretching and progressive exercises, plus scapular taping Complete evaluations at baseline, mid-program, and after the program, including goniometry (ROM), manual muscle testing, pain scale (VAS), postural assessment, and a functional ability checklist

DETAILED DESCRIPTION:
This study is a single-patient case report describing the design, delivery, and observed response to a pre-operative rehabilitation program for a pediatric patient with deformity involving the humeral head and shaft. The report will document the patient's baseline presentation, the clinical reasoning used to select pre-operative rehabilitation goals, and the step-by-step rehabilitation approach used to optimize the shoulder and upper-limb condition before planned surgical management.

The rehabilitation program is intended to maximize safe functional capacity pre-operatively by addressing modifiable impairments commonly associated with this condition, such as pain, limited range of motion, weakness, altered scapulohumeral mechanics, and compensatory movement patterns. The case report will describe treatment components (e.g., education, therapeutic exercise, flexibility and strengthening strategies, neuromuscular re-education, and other noninvasive physical therapy modalities as clinically indicated), how the program is progressed over time, and any precautions used to ensure age-appropriate and condition-appropriate care.

To evaluate response to the program, the study will collect structured pre- and post-program measurements relevant to shoulder/upper-limb status, such as:

* Pain and symptom severity
* Shoulder range of motion
* Muscle strength and/or functional performance
* Activity limitations and functional use of the affected arm
* Observed posture and movement quality (as clinically applicable) The report will also capture treatment adherence, any adverse events, and notable barriers/facilitators to participation (e.g., tolerance, fatigue, caregiver involvement). Findings will be presented descriptively to help clinicians and families understand what a pre-operative rehabilitation plan may include for a child with humeral deformity, and what types of short-term changes may be observed during the pre-surgical period.

ELIGIBILITY:
Inclusion Criteria:

- Not applicable (case report; single patient case).

Exclusion Criteria:

- Not applicable (case report; single patient case).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Range of Motion | 4 weeks
  Shoulder range of motion will be assessed using a standard universal goniometer to quantify the motion of the affected upper limb.
Manual Muscle Testing | 4 weeks
  Upper-limb and shoulder muscle strength will be assessed using standardized Manual Muscle Testing procedures. Key muscle groups around the shoulder and scapula (e.g., shoulder flexors, abductors, internal/external rotators, and scapular stabilizers)
Functional Ability | 4 weeks
  Functional status of the affected upper limb will be assessed using the Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) questionnaire. The patient (with caregiver assistance as needed) will rate the difficulty of performing common daily activities and the impact of symptoms such as pain on function. Responses are summed and converted to a 0-100 score, where higher scores indicate greater disability.

SECONDARY OUTCOMES:
Pain intensity | 4 weeks
  Pain intensity will be measured using a Visual Analog Scale (VAS). The patient will be asked to rate her pain by marking on a 10-cm line anchored by "no pain" (0) and "worst pain imaginable" (10).

CONTACTS AND LOCATIONS:
Locations (1):
- Out patinets clinics, Faculty of Physical Therapy Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No